CLINICAL TRIAL: NCT00854594
Title: Interprofessional Training for Improving Diabetes Care
Brief Title: Interprofessional Training to Improve Diabetes Care: The ReSPECT Trial
Acronym: ReSPECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Case Western Reserve University (Other); The Cleveland Clinic (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EDU 08-414
Record Dates: First submitted 2009-02-27; First posted 2009-03-03 (Estimated); Results first posted 2015-10-06 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-09

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes; Telemedicine; Shared Medical Appointments
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Control sites will receive the baseline measures pre and post. These sites will receive traditional diabetes education, which includes teleconsultation.
- ReSPECT Intervention (Experimental): Intervention sites will receive baseline measures pre and post, but also in-depth Shared Medical Appointments (SMA)(The Role modeling in Shared medical appointments to Promote Establishing Collaborative Teams (ReSPECT) intervention) and at 15 months SMA video conferences. At the end of the 18 months the randomly selected patients and providers will be asked to take part in a qualitative interview.
  Interventions: Behavioral: Role modeling in Shared medical appointments to Promote Establishing Collaborative Teams (ReSPECT)

INTERVENTIONS:
Behavioral: Role modeling in Shared medical appointments to Promote Establishing Collaborative Teams (ReSPECT) — The intervention is designed to educate the clinicians at intervention CBOCs by modeling interprofessional team practices during SMAs for diabetes mellitus (DM) patients from each CBOC primary care provider's (PCP) patient panel. We hypothesize that this education at intervention CBOCs will improve interprofessional practices and overall quality care delivered to veterans.
  Other Names: ReSPECT
  Arms: ReSPECT Intervention

SUMMARY:
The investigators' study focuses on improving the care of diabetes, a complex chronic illness, by providing important insights into interprofessional training and its potential role in fostering the necessary interdisciplinary management needed for chronic conditions and in addressing the gap between best practice and actual care provided.

DETAILED DESCRIPTION:
The complexity of diabetes management challenges the acute care-oriented healthcare system. Some experts suggest part of the problem is that the healthcare system fosters a separate silos decision making model. While there is increasing recognition that quality diabetes care is best provided in an interdisciplinary manner, interprofessional training models are limited, as is understanding of the links between interprofessional training, actual practice, and patient outcomes. Advancing our understanding of interprofessional training models is critical because most of the complications associated with diabetes (e.g., amputations, renal failure, strokes) can be prevented or delayed with proper management. The investigators' objective is to better understand the processes and mechanisms by which interprofessional training impacts on chronic care management (practice patterns) and the ways it translates into improved patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

CLINICIANS

* All clinicians in all of Ohio's CBOCs (except for the Georgetown CBOC) will be eligible for the study (all PCPs have patients with DM in their panel of patients).

PATIENTS

* All diabetic patients who are seen in Ohio's CBOCs (except for the Georgetown CBOC) will be eligible for the study.

Exclusion Criteria:

CLINICIANS

* Any clinician who does not have diabetic patients on their panel, who aren't apart of Ohio's CBOC's, or see patients at the Georgetown CBOC will not be eligible to participate.

PATIENTS

* Patients who don't have a diagnosis of diabetes, who aren't seen at one of Ohio's CBOC's, or is seen for their medical care at the Georgetown CBOC will not be eligible to participate.

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2010-09; Primary Completion 2013-05 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan R Kirsh, MD, Principal Investigator — HSR&D Central Office
Locations (1):
- Louis Stokes VA Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Result] Kirsh SR, Schaub K, Aron DC. Shared medical appointments: a potential venue for education in interprofessional care. Qual Manag Health Care. 2009 Jul-Sep;18(3):217-24. doi: 10.1097/QMH.0b013e3181aea27d. PMID 19609192

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Cleveland and Cincinnati CBOCs (excluding Georgetown; n = 18 CBOCs) were the study sites randomized to the two study arms. Providers within site were subject to the intervention to which the site was randomized and the questionnaire responses were collected at the provider level.
Groups:
- Control: Providers within sites randomized to the control arm will receive the baseline measures pre and post. These sites will receive traditional diabetes education, which includes teleconsultation.
- ReSPECT Intervention: Providers within sites randomized to the intervention arm will receive baseline measures pre and post, but also in-depth Shared Medical Appointments (SMA)(The Role modeling in Shared medical appointments to Promote Establishing Collaborative Teams (ReSPECT) intervention) and at 15 months SMA video conferences. At the end of the 18 months the randomly selected patients and providers will be asked to take part in a qualitative interview.
  Role modeling in Shared medical appointments to Promote Establishing Collaborative Teams (ReSPECT): The intervention is designed to educate the clinicians at intervention Community-Based Outpatient Clinics (CBOCs) by modeling interprofessional team practices during SMAs for diabetes mellitus (DM) patients from each CBOC primary care provider's (PCP) patient panel. We hypothesize that this education at intervention CBOCs will improve interprofessional practices and overall quality care delivered to veterans.
Period: Overall Study
Arm/Group | Control | ReSPECT Intervention
Started | 48 (9 sites randomized to control arm, providers completed surveys before and/or after study period) | 69 (9 sites randomized to intervention, providers completed surveys before and/or after study period)
Completed | 48 | 69
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: For providers who completed the survey once, using demographics reported; for providers who completed the survey twice, using demographics from earlier survey completion.
Groups:
- ReSPECT Intervention: Intervention sites will receive baseline measures pre and post, but also in-depth Shared Medical Appointments (SMA)(The Role modeling in Shared medical appointments to Promote Establishing Collaborative Teams (ReSPECT) intervention) and at 15 months SMA video conferences. At the end of the 18 months the randomly selected patients and providers will be asked to take part in a qualitative interview.
  Role modeling in Shared medical appointments to Promote Establishing Collaborative Teams (ReSPECT): The intervention is designed to educate the clinicians at intervention CBOCs by modeling interprofessional team practices during SMAs for DM patients from each CBOC primary care provider's (PCP) patient panel. We hypothesize that this education at intervention CBOCs will improve interprofessional practices and overall quality care delivered to veterans.
- Total: Total of all reporting groups
Arm/Group | Control | ReSPECT Intervention | Total
Number analyzed (Participants) | 48 | 69 | 117
Age, Customized [Number; unit: participants] — Age categories indicated in provider questionnaire.
  participants
    Missing | 0 | 4 | 4
    39 years or less | 7 | 12 | 19
    40 to 59 years | 41 | 48 | 89
    60 years or greater | 0 | 5 | 5
Sex/Gender, Customized [Number; unit: participants]
  Male | 12 | 13 | 25
  Female | 36 | 53 | 89
  Unknown | 0 | 3 | 3

OUTCOME MEASURES:

1. Secondary Outcome: Attitudes Toward Healthcare Teams Scale and Subscales
Description: A validated scale developed to assess attitudes towards teams in a healthcare setting with three subscales to assess attitudes toward team value, attitudes toward team efficiency, and attitudes towards physician's shared role on a team. Each of the 21 items is rated 1 to 6, ranging from 'Strongly Disagree' to 'Strongly Agree'. The scale was considered 'complete' for analysis among providers who answered at least 7 of the 21 items. Items were reverse-coded as specified in the subscale development publication. Averages across completed items were calculated within provider. Higher values corresponded with more positive attitudes towards teams.
Time Frame: Baseline
Population: Providers within sites randomized to control and intervention arms were surveyed at baseline; 39 control arm providers and 53 intervention arm providers complete the attitude scale of the survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | ReSPECT Intervention
Number analyzed (Participants) | 39 | 53
units on a scale | 4.42 (.52) | 4.29 (.55)

2. Primary Outcome: Provider Abilities Scale - Subscale From the Midwest (MW) Clinicians' Network
Description: Providers asked to indicate their level of confidence on an 11-point scale, with 0 indicating 'not at all confident' and 10 indicating 'extremely confident' for the following activities:
  1. Instruct patients on home glucose monitoring
  2. Teach foot care
  3. Teach insulin administration
  4. Instruct patients about diet
  5. Help patients make changes in their diets that you have recommended
  6. Instruct patients about regular exercise
  7. Help patients make changes in their exercise habits that you have recommended
  8. Identify candidates for long-acting insulin
  9. Interpret glucose patterns
  10. Adjust insulin in insulin-treated patients with poor glycemic control
  11. Do you feel comfortable knowing whether to titrate basal insulin versus bolus insulin
  12. Manage patients with poor glycemic control
  13. Initiate insulin therapy (NPH or insulin glargine and aspart)
  14. Apply principles of diabetes care in a team setting
  Averages of provider efficacy were calculated across all activities.
Time Frame: Baseline
Population: Providers within sites randomized to control and intervention arms were surveyed at baseline; 39 control arm providers and 55 intervention arm providers completed the ability items of the survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | ReSPECT Intervention
Number analyzed (Participants) | 39 | 55
units on a scale | 6.89 (2.17) | 6.41 (1.90)
Statistical Analysis 1: Comparison: Control vs ReSPECT Intervention; Null hypothesis: pre-intervention efficacies will be equal in the two study arms; Test type: Superiority or Other; p = 0.26, t-test, 2 sided

3. Primary Outcome: Provider Abilities Scale - Subscale From the Midwest (MW) Clinicians' Network
Description: as for outcome 2
Time Frame: 22 months (post-intervention)
Population: Providers within sites randomized to control and intervention arms were surveyed after the intervention period; 20 control arm providers and 29 intervention arm providers completed the ability items of the survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | ReSPECT Intervention
Number analyzed (Participants) | 20 | 29
units on a scale | 7.09 (2.05) | 6.88 (2.14)
Statistical Analysis 1: Comparison: Control vs ReSPECT Intervention; Null hypothesis: post-intervention efficacies will be equal in the two study arms; Test type: Superiority or Other; p = 0.74, t-test, 2 sided

4. Secondary Outcome: Attitudes Toward Healthcare Teams Scale and Subscales
Description: as for outcome 1
Time Frame: 22 months (post-intervention)
Population: Providers within sites randomized to control and intervention arms were surveyed after the intervention period; 20 control arm providers and 29 intervention arm providers completed the attitude scale of the survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | ReSPECT Intervention
Number analyzed (Participants) | 20 | 29
units on a scale | 4.44 (0.52) | 4.24 (0.59)

ADVERSE EVENTS:
Arm/Group | Control | ReSPECT Intervention
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/69
Other Adverse Events (participants affected / at risk) | 0/48 | 0/69

LIMITATIONS AND CAVEATS:
IRB-related delays were so significant that aspects of the research plan could not be completed. Delays have also been experienced in the collection and analysis of clinical endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes